CLINICAL TRIAL: NCT02770430
Title: A Phase II, Randomized Study to Evaluate the Human Mesenchymal Stem Cells as a First-line Treatment for aGVHD in Patients Steroids Resistant.
Brief Title: Mesenchymal Stem Cells as First Treatment Line for Resistant Acute Graft Versus Host Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 12-0407
Record Dates: First submitted 2015-10-08; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Graft vs Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional treatment (Active Comparator): After randomization, patients will be allocated to receive conventional treatment:
  1. Basiliximab 20mg dose for adults and 10mg for children, 1 time a week or every 3 days if worsens the stage of GVHD until reaching Very Good Partial Response (VGPR) or for a maximum of 4 doses, whichever comes first.
  2. If after the item (1) will not obtained VGPR: Infliximab 5 to 10 mg/kg dose, 1 time a week, four weeks or even VGPR.
  Interventions: Drug: conventional treatment
- mesenchymal stem cells (Experimental): Patients in the study group will receive two infusions of MSC per week during two weeks and 1 more MSC infusion (2 + 2 + 1 scheme). Dosage: 2x10E6/Kg
  Interventions: Biological: mesenchymal stem cells

INTERVENTIONS:
Biological: mesenchymal stem cells — MSCs derived from bone marrow (BM) will be isolated and expanded in the laboratory under conditions of Good Manufacturing Practice. The quality control involves immunophenotyping, differentiation, microbiological control, mycoplasma and endotoxin tests. Patients will receive five infusions of MSC. Dosage: 2x10E6 cells/Kg
  Other Names: mesenchymal stomal cells
  Arms: mesenchymal stem cells
Drug: conventional treatment — 1. Basiliximab 20mg dose for adults and 10mg for children, 1 time a week or every 3 days if worsens the stage of GVHD until reaching Very Good Partial Response (VGPR) or for a maximum of 4 doses, whichever comes first.
  2. If after the item (1) will not obtained VGPR: Infliximab 5 to 10 mg/kg dose, 1 time a week, four weeks or even VGPR.
  Other Names: Basiliximab and/or Infliximab
  Arms: conventional treatment

SUMMARY:
Steroids are still the first line treatment for established severe acute-graft-versus-host-disease (aGVHD), with a response rate of 30-50%, and there is no established and effective therapy for severe steroid-refractory (aGVHD). The outcome for patients is poor and overall survival low, with few patients alive at 2 years.

In the case of failure after corticosteroid treatment, different therapeutic options have been introduced as second or third-line strategies. In this scenario, infusion of ex vivo expanded mesenchymal stromal cells (MSCs) has emerged as an additional tool for treatment of GVHD.

The purpose of this work is conduct a study in patients with refractory and/or resistant GVHD corticosteroids treatment. It will be randomized into two groups: one group that will receive the MSCs and the other group will follow the acute GVHD steroid-resistant and/or refractory treatment according to the routines of the Bone Marrow Transplantation (BMT) service of Hospital de Clinicas de Porto Alegre. It will be evaluated aspects of immune recovery early after MSCs infusion.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplant (AlloSCT) is the treatment of choice for many malignant and non-malignant hematological disorders. However, this treatment is frequently complicated by acute graft-versus-host-disease (aGVHD), wich can be associated with high morbidity and mortality.

Steroids are still the first line treatment for established aGVHD, with a response rate of 30-50%, and there is no established and effective therapy for severe steroid-refractory aGVHD. The outcome for patients is poor and overall survival low, with few patients alive at 2 years.

In the case of failure after corticosteroid treatment, different therapeutic options have been introduced as second or third-line strategies. In this scenario, infusion of ex vivo expanded mesenchymal stem cells (MSCs) has emerged as an additional tool for treatment of GVHD.

MSCs are non hematopoietic multipotent cells with self-renewal properties and the ability to differentiate into mesenchymal tissues. Several lines of evidence in the past few years have confirmed the ability of theses cells differentiate into cells derived form embryonic mesoderm, such as osteocytes, adipocytes and chondroblasts. In vitro, culture-expanded MSCs express membrane antigens that can be immunophenotyped by flow cytometry. The most widely accepted antigen expression pattern is cluster of differentiation (CD) 29, CD105, CD73, and CD90 positivity in 97 % of cells and minimal expression of CD45, CD34, CD3, CD14, CD19, or human leukocyte antigen (HLA) -DR, which should be positive in less than 3 % of cells.

Because they are easy to isolate and culture and due to their differentiation potential and production of growth factors and cytokines, MSC have become ideal candidates for regenerative protocols.

The purpose of this work is conduct a study in patients with refractory and/or resistant GVHD corticosteroids treatment. It will be randomized into two groups: one group that will receive the MSCs and the other group will follow the acute GVHD steroid-resistant and/or refractory treatment according to the routines of the Bone Marrow Transplantation service of Hospital de Clinicas de Porto Alegre. It will be evaluated aspects of immune recovery early after MSCs infusion.

METHOD: This is a prospective, randomized, controlled, open label study to evaluate the effectiveness of early treatment of steroid-resistant acute GVHD with MSC. All patients with refractory and/or resistant steroids GVHD will be included after signing of free and informed consent.

After randomization, patients will be allocated to receive conventional treatment:

1. Basiliximab 20mg dose for adults and 10mg for children, 1 time a week or every 3 days if worsens the stage of GVHD until reaching Very Good Partial Response (VGPR) or for a maximum of 4 doses, whichever comes first.
2. If after the item (1) will not obtained VGPR: Infliximab 5 to 10 mg/kg dose, 1 time a week, four weeks or even VGPR.

Patients in the study group will receive two infusions of MSC per week during two weeks and 1 more MSC infusion (2 + 2 + 1 scheme).

After 28 days, if VGPR is not obtained, crossover between groups will be allowed as well as for the patients with progressive GVHD in spit of treatment arm, before day +28. The latter group of patients, who use both treatments (MSC + Conventional treatment) before day + 28 will be analyzed separately.

Bone marrow (BM) derived MSCs from normal BMT donors (third part) will be isolated and expanded under conditions of Good Manufacturing Practice. The quality control involves immunophenotyping, differentiation, microbiological control, mycoplasma and endotoxin tests.

Patients response evaluation will be at Day + 28:

1. Complete response: disappearance of all symptoms
2. Partial response: with a decrease at least of one degree of GVHD
3. VGPR: decrease to the stage I of GVHD
4. Stable disease: when there is a stability of the disease
5. Number and type of infection in the first 100 days after transplant

The transplant-related mortality, disease-free survival, overall survival and the development of chronic GVHD or not, will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* All patients with refractory and/or resistant steroids GVHD will be included after signing of free and informed consent.

Exclusion Criteria:

* They will be excluded from the study, patients who did not agree to participate and don't sign an informed consent (which is going to receive conventional treatment) and that patients who is a Grade I refractory GVHD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Complete response: disappearance of all symptoms | It will be evaluated the patients response who received MSC infusion or conventional therapy in the 28th day of the study.

SECONDARY OUTCOMES:
Partial response: with a decrease at least of one degree of GVHD | It will be evaluated the patients response who received MSC infusion or conventional therapy in the 28th day of the study.
VGPR: decrease to the stage I of GVHD | It will be evaluated the patients response who received MSC infusion or conventional therapy in the 28th day of the study.
Stable disease: when there is a stability of the disease (by Clinical evaluation) | It will be evaluated the patients response who received MSC infusion or conventional therapy in the 28th day of the study.
Number of infection (by Clinical and laboratory evaluation) | First 100 days after transplant
Type of infection (by Clinical and laboratory evaluation) | First 100 days after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Lucia S Silla, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Centro Terapia e Tecnologia Celular, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided